CLINICAL TRIAL: NCT02805101
Title: A Comparative Study of the Performance of Biodentine and Mineral Trioxide Aggregate (MTA) in Sealing Root Perforations.
Brief Title: Comparative Study Between Biodentine and Mineral Trioxide Aggregate in Sealing Root Perforations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-OperDent-02-2016
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Root Perforation at the Bifurcation Area
MeSH Terms: interventions — tricalcium silicate; Pemetrexed

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biodentine (Experimental): The perforation area of the root is going to be covered by Biodentine
  Interventions: Drug: Biodentine
- MTA (Active Comparator): The perforation area of the root is going to be covered by MTA.
  Interventions: Drug: MTA

INTERVENTIONS:
Drug: Biodentine — Biodentine is going to be used as the sealing agent for the perforation.
  Arms: Biodentine
Drug: MTA — MTA is going to be used as the sealing agent for the perforation.
  Arms: MTA

SUMMARY:
This is a study aimed to compare two materials: (1) Biodentine and (2) MTA. These two materials are going to be tested in sealing accidental root perforations at the bifurcation areas. The study is going to be conducted as a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. vital molars (upper or lower )
2. suffered from perforation in the bifurcation area of the roots through a process of open access cavity, taking into account the location and size of perforation
3. Perforation should not exceed the size of 3 mm
4. Perforation and must also take into account the time of perforation.

Exclusion Criteria:

1. If the molar not vital.
2. If the perforation not in bifurcation root or extended inside the canals.
3. Size of perforation larger than 3 mm.
4. A long time ago on the occurrence of perforation with resorption in tooth structure.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2017-06-20 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Success at 3 months following root sealing | The success of treatment is assessed at three months following the application of the material
  Case is considered successful if clinical and radiographic examinations of the tooth are sound 100%.
Success at 6 months following root sealing | The success of treatment is assessed at 6 months following the application of the material
  Case is considered successful if clinical and radiographic examinations of the tooth are sound 100%.
Success at 9 months following root sealing | The success of treatment is assessed at 9 months following the application of the material
  Case is considered successful if clinical and radiographic examinations of the tooth are sound 100%.
Success at 12 months following root sealing | The success of treatment is assessed at 12 months following the application of the material
  Case is considered successful if clinical and radiographic examinations of the tooth are sound 100%.
Success at 18 months following root sealing | The success of treatment is assessed at 18 months following the application of the material
  Case is considered successful if clinical and radiographic examinations of the tooth are sound 100%.
Success at 24 months following root sealing | The success of treatment is assessed at 24 months following the application of the material
  Case is considered successful if clinical and radiographic examinations of the tooth are sound 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad MN Aldakak, DDS MSc, Principal Investigator — PhD Student in Operative Dentistry; Souad Abboud, DDS MSc PhD, Study Chair — Associate Professor of Operative Dentistry, University of Damascus Dental School, Damascus, Syria
Locations (1):
- Department of Operative Dentistry, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guneser MB, Akbulut MB, Eldeniz AU. Effect of various endodontic irrigants on the push-out bond strength of biodentine and conventional root perforation repair materials. J Endod. 2013 Mar;39(3):380-4. doi: 10.1016/j.joen.2012.11.033. Epub 2013 Jan 16. PMID 23402511
- [Background] Iwamoto CE, Adachi E, Pameijer CH, Barnes D, Romberg EE, Jefferies S. Clinical and histological evaluation of white ProRoot MTA in direct pulp capping. Am J Dent. 2006 Apr;19(2):85-90. PMID 16764130
- [Background] Koubi G, Colon P, Franquin JC, Hartmann A, Richard G, Faure MO, Lambert G. Clinical evaluation of the performance and safety of a new dentine substitute, Biodentine, in the restoration of posterior teeth - a prospective study. Clin Oral Investig. 2013 Jan;17(1):243-9. doi: 10.1007/s00784-012-0701-9. Epub 2012 Mar 14. PMID 22411260
- [Background] Laurent P, Camps J, De Meo M, Dejou J, About I. Induction of specific cell responses to a Ca(3)SiO(5)-based posterior restorative material. Dent Mater. 2008 Nov;24(11):1486-94. doi: 10.1016/j.dental.2008.02.020. Epub 2008 Apr 29. PMID 18448160
- [Background] Zanini M, Sautier JM, Berdal A, Simon S. Biodentine induces immortalized murine pulp cell differentiation into odontoblast-like cells and stimulates biomineralization. J Endod. 2012 Sep;38(9):1220-6. doi: 10.1016/j.joen.2012.04.018. Epub 2012 Jul 24. PMID 22892739